CLINICAL TRIAL: NCT06198582
Title: Evaluation of the Effect of Virtual Reality Based Task Specific Exercises on Functional Level and Disease Related Quality of Life in Patients With Hand Flexor Tendon Injury
Brief Title: The Effect of Virtual Reality Based Task Specific Exercises in Patients With Hand Flexor Tendon Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mert Karacay, Physical Medicine and Rehabilitation Resident, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 263799996/75
Record Dates: First submitted 2023-11-21; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Tendon Injury - Hand; Flexor Tendon Rupture
Keywords: flexor tendon rehabilitation; virtual reality; task specific exercise
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention Group (Experimental): Consisted of patients who received a virtual reality-based task-specific exercise programme in addition to the early passive mobilisation programme
  Interventions: Other: Virtual Reality Exercises
- Control Group (No Intervention): Consisted of patients who received the early passive mobilisation programme

INTERVENTIONS:
Other: Virtual Reality Exercises — In addition to conventional treatment, patients in the study group underwent a virtual reality-based task-specific exercise program in a computer-based virtual reality station. Two different virtual reality games that fit the definition of task-specific exercise were selected for our study. In order for the patient to complete the task in the game, the patient was asked to extend the upper extremity and hand to touch the virtual object through the reflection on the screen and to first grasp the object in the virtual environment by making active flexion with all fingers and to move it from one place to another on a certain plane without disturbing the grasping posture of the hand. These virtual reality exercises selected in our study were practiced under the supervision of the researcher 3 days a week for 15 minutes each for a total of 4 weeks. These sessions consisted of three sets of 2.5 minutes each for each game, with 15-second breaks between sets.
  Arms: Virtual Reality Intervention Group

SUMMARY:
This study,the investigators aimed to investigate the effects of virtual reality-based task-specific exercises applied in addition to conventional rehabilitation program on functional level and disease-related quality of life in patients who underwent surgical repair due to flexor tendon damage due to traumatic hand injury.

ELIGIBILITY:
Inclusion Criteria:

* Tendon repair operation due to flexor tendon injury in one hand
* Admission to the Traumatic Hand Rehabilitation Outpatient Clinic of Ankara City Hospital Physical Medicine and Rehabilitation Hospital within the first postoperative week and enrolled in an early passive mobilization program
* Must be in the sixth post operative week

Exclusion Criteria:

* Under 18 years of age
* Concomitant extensor tendon injury
* Having any accompanying orthopedic, neurologic, rheumatologic and vascular problems in the premorbid period
* Presence of cognitive deficit
* Presence of visual field deficit
* Presence of postural instability
* Presence of epilepsy and/or cyber disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in short form-36 (SF-36) scores | Pre-intervention (postoperative sixth week), immediately after the intervention (postoperative tenth week)
  A scale used for determining quality of life. This form evaluates the quality of life under 9 different headings. Minimum value of all headings is %0 and maximum is %100. Higher scores mean a better outcome.
The functional level of dexterity and coordination | Pre-intervention (postoperative sixth week), immediately after the intervention (postoperative tenth week)
  The functional level of dexterity and coordination was assessed with the Nine-Hole Peg Test. The test material for this test consists of nine standardised pegs and a board with nine holes equidistant from each other. When the patient feels ready, the patient is asked to close the nine holes as quickly as possible, regardless of the order of the sticks, provided that the patient places one stick at a time. Once all the holes have been filled, without a break, the patient is asked to remove the rods one by one from the holes and put them back where they came from. From the moment the patient touches the first stick, the observer starts timing. When the last rod is removed and placed in the area where the rods were taken, the time is stopped and recorded. In measurements made in different periods in the same patient, completion of the test in a shorter time indicates improvement in hand skills.
Dexterity-related activity limitations in activities of daily living | Pre-intervention (postoperative sixth week), immediately after the intervention (postoperative tenth week)
  Dexterity-related activity limitations in activities of daily living were assessed by Duruöz hand index and Quick Disability of Arm, Shoulder and Hand. Duruöz hand index includes 18 questions on manual dexterity related to "kitchen work, dressing, personal hygiene, office work and other activities of daily living". The questionnaire takes approximately 2-3 minutes to complete. The minimum score that can be obtained from the questionnaire is 0 points while the maximum score is 90 points. A lower score indicates fewer limitations in activities of daily living. The Quick Arm, Shoulder and Hand Disability Scale consists of 11 questions. Minimum value of the scale is 0 and maximum is 100. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Grip strength | Pre-intervention (postoperative sixth week), immediately after the intervention (postoperative tenth week)
  The grip strength was measured with a Jamar dynamometer. The measured value was recorded in kilograms.
Change in active range of motion | Pre-intervention (postoperative sixth week), immediately after the intervention (postoperative tenth week)
  Range of motion was measured using a standard hand goniometer and the measured degree was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)